CLINICAL TRIAL: NCT00280800
Title: Effectiveness of Auto-adjusted Continuous Positive Airway Pressure for Long-term Treatment of Obstructive Sleep Apnea Syndrome
Brief Title: Effectiveness of Auto-adjusted Continuous Positive Airway Pressure for Long-term Treatment of Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konrad E. Bloch (Other)
Collaborators: University of Zurich (Other); Kantonsspital Münsterlingen (Other); Zuercher Hoehenklinik Wald (Other); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor-Investigator, Konrad E. Bloch, Professor, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EK 1187
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: randomized; controlled; double blind; effectiveness; auto CPAP; treatment; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): constant CPAP
  Interventions: Device: constant CPAP devices
- 2 (Experimental): automatic CPAP
  Interventions: Device: automatic CPAP devices

INTERVENTIONS:
Device: constant CPAP devices — different CPAP mode
  Arms: 1
Device: automatic CPAP devices — different CPAP mode
  Arms: 2

SUMMARY:
Hypothesis: Computer controlled continuous positive airway pressure (autoCPAP) is equally effective in improving obstructive sleep apnea syndrome symptoms, breathing disturbances, objective vigilance, and it is cost-effective compared to conventional fixed continuous positive airway pressure.

DETAILED DESCRIPTION:
1. To investigate whether computer controlled continuous positive airway pressure (autoCPAP) improves subjective sleepiness, quality of life, objective vigilance, and nocturnal respiration to a similar degree as conventional fixed continuous positive airway pressure in the initial phase of treatment and over the subsequent 2 years during home therapy
2. To investigate the cost of autoCPAP compared to fixed CPAP therapy

ELIGIBILITY:
Inclusion Criteria:

* Excessive sleepiness, and Epworth Sleepiness Score > or = 8
* Apnea- Hypopnea-Index (AHI) > or = 10/hour
* Age 18-75

Exclusion Criteria:

* Psychophysiological incapacity to perform questionnaires
* Other sleep disorders
* Psychiatric disease requiring treatment
* Previous CPAP therapy
* Previous uvulopalatopharyngoplasty
* Chronic nasal obstruction that required treatment for more than 1 month
* Cancer
* COPD, with FEV1 < 50% predicted
* Symptomatic cardiovascular disease requiring treatment defined as congestive heart failure > NYHA II
* Previous stroke with neurological residuum
* Cheyne-Stokes respiration
* Chronic pain syndromes, fibromyalgia
* Drug or alcohol addiction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2006-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
subjective sleepiness and other OSAS symptoms | 3 months, 1 year, 2 years
quality of life | 3 months, 1 year, 2 years
percentage of withdrawal and cross-over to other CPAP mode | 3 months, 1 year, 2 years
objective vigilance | 3 months, 1 year, 2 years
blood pressure | 3 months, 1 year, 2 years
cost/utility ratios | 3 months, 1 year, 2 years

SECONDARY OUTCOMES:
major outcomes in subgroups of patients with severe and mild OSAS | 3 months, 1 year, 2 years
circulating markers of inflammation and cardiovascular risk | 3 months, 1 year, 2 years
side effects | 3 months, 1 year, 2 years
nocturnal respiratory disturbances | 3 months, 1 year, 2 years
treatment adherence | 3 months, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — Pulmonary Division and Sleep Disorders Center, University Hospital of Zürich, Switzerland
Locations (1):
- Pulmonary Division and Sleep Disorders Center, University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Crook S, Sievi NA, Bloch KE, Stradling JR, Frei A, Puhan MA, Kohler M. Minimum important difference of the Epworth Sleepiness Scale in obstructive sleep apnoea: estimation from three randomised controlled trials. Thorax. 2019 Apr;74(4):390-396. doi: 10.1136/thoraxjnl-2018-211959. Epub 2018 Aug 12. PMID 30100576
- [Derived] Bloch KE, Huber F, Furian M, Latshang TD, Lo Cascio CM, Nussbaumer-Ochsner Y, Senn O, Russi EW, Kohler M, Schoch OD, Turk A, Imhof E, Laube I, Matthews F, Thurnheer R. Autoadjusted versus fixed CPAP for obstructive sleep apnoea: a multicentre, randomised equivalence trial. Thorax. 2018 Feb;73(2):174-184. doi: 10.1136/thoraxjnl-2016-209699. Epub 2017 Oct 5. PMID 28982804
- See also: Bloch KE et al. Thorax 2017;0:1-11 — http://www.ncbi.nlm.nih.gov/pubmed/?term=28982804
- See also: Link to publication — http://dx.doi.org/10.1136/thoraxjnl-2016-209699